CLINICAL TRIAL: NCT00274391
Title: Efficacy of Amiloride and Hypertonic Saline in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DONALDS00A0
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2006-01-10 (Estimated); Status verified 2005-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Amiloride

INTERVENTIONS:
Drug: 7% NaCl
Drug: Amiloride HCl

SUMMARY:
The purpose of this research study is to determine whether the combination of inhaled amiloride and a concentrated salt solution is better than the salt solution itself for cystic fibrosis (CF) patients. In CF, airway secretions are thick and dehydrated. Many patients use inhaled salt solutions to help draw water into their secretions so that they are easier to get rid of with chest physiotherapy ("chest PT") and cough. Unfortunately, these salt solutions are reabsorbed very quickly by the airways, so the beneficial effects may not last very long. In the hopes of prolonging their effects, the drug amiloride could be used in combination to slow salt and water reabsorption from airways. Amiloride is a medication that has been given by mouth for high blood pressure for many years. It is possible that the combination of salt solutions and inhaled amiloride may significantly improve the clearance of secretions in CF, which would be expected to improve lung function in CF.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CF
* 2 gene mutations identified, or
* Sweat chloride > 60 mmol/L, and
* 1 or more typical CF clinical features
* Age > 14 years
* Able to perform spirometry and have post-bronchodilator FEV1 > 50% of predicted at screening
* Oxyhemoglobin saturation (by pulse oximetry) > 92% on room air
* Able to provide informed consent

Exclusion Criteria:

* Unstable lung disease:
* FEV1 > 15% below best clinical measurement within 6 months
* Requirement for IV antibiotics within 4 weeks of screening
* Requirement for any change in pulmonary medication within 2 weeks of screening
* Evidence of reactive airways
* Clinical diagnosis of asthma

  -> 15% increase in FEV1 after bronchodilator at screening
* Hypertonic saline use within 2 weeks of screening
* Unwilling or unable to either continue or discontinue cyclical therapies (e.g. inhaled tobramycin) for the 2 weeks prior to screening and the entire study period
* Pregnancy, breast-feeding, or unwillingness to use barrier contraception during the entire study period
* History of allergy or intolerance to amiloride, hypertonic saline, quinine, albuterol, or related compounds
* Renal insufficiency (creatinine > 1.5 mg/dl)
* Hyperkalemia (K+ > 5.0 meq/L)
* Investigational drug use within 30 days of screening
* Radiation exposure within the past year that would exceed Federal Regulations by participating in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2001-07; Study Completion 2004-04

PRIMARY OUTCOMES:
FEV1

SECONDARY OUTCOMES:
Mucociliary clearance rate
Quality of Life
FVC
FEF25-75
Cough clearance rate

CONTACTS AND LOCATIONS:
Overall Officials: Scott H. Donaldson, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States